CLINICAL TRIAL: NCT05384769
Title: Feasibility Study of Lung Cancer Screening Using Cell-Free DNA Liquid Biopsy at Home in High-Risk Current and Former Smokers
Brief Title: Feasibility of Cell-Free DNA Liquid Biopsy in Screening High-Risk Patients for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21591; NCI-2022-02513 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21591 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-04-19; First posted 2022-05-20 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (liquid biopsy, optional LDCT) (Experimental): Participants undergo collection of blood sample (liquid biopsy), with option to undergo LDCT if liquid biopsy results are positive.
  Interventions: Procedure: Liquid Biopsy; Procedure: Low Dose Computed Tomography of the Chest; Other: Survey Administration
- Cohort B (LDCT, optional liquid biopsy) (Experimental): Participants undergo low dose CT with optional liquid biopsy on the same day as LDCT.
  Interventions: Procedure: Liquid Biopsy; Procedure: Low Dose Computed Tomography of the Chest; Other: Survey Administration

INTERVENTIONS:
Procedure: Liquid Biopsy — Undergo liquid biopsy
  Other Names: Plasma Biopsy
Procedure: Low Dose Computed Tomography of the Chest — Undergo low dose CT
  Other Names: LDCT; Low Dose Chest Computed Tomography; Low-dose Chest Computed Tomography; Low-dose Chest CT
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial investigates how practical and doable (feasibility) cell-free deoxyribonucleic acid (DNA) liquid biopsy is in screening high-risk patients for lung cancer. Currently, a low dose computed tomography (CT) scan is used to screen for lung cancer, however, due to various factors, few high-risk patients are screened. Liquid biopsy utilizes technology that can detect small amounts of DNA shed by cancer cells and may be able to spot lung cancer at an earlier stage. If a positive result comes back from the liquid biopsy, a patient may be more willing to get a low dose CT (LDCT) scan, possibly confirming the biopsy's findings and thus leading to more early lung cancer detection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of lung cancer screening using liquid biopsy in a community setting.

SECONDARY OBJECTIVES:

I. To determine screening follow-through rates in those who agreed to undergo screening by preferred modality (liquid biopsy versus [vs] LDCT).

II. To determine the rate of LDCT following liquid biopsy (in those who underwent liquid biopsy) after stratifying by test result (negative versus positive).

III. To compare participant sociodemographic factors (age, sex, race/ethnicity, educational background) and survey scores across screening preference (liquid biopsy vs. LDCT).

OUTLINE: Participants choose 1 of 2 cohorts.

COHORT A: Participants undergo collection of blood sample (liquid biopsy), with option to undergo LDCT if liquid biopsy results are positive.

COHORT B: Participants undergo low dose CT with optional liquid biopsy on the same day as LDCT.

After completion of study, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented written informed consent of the participant.
* Age 50-80 years.
* Smoking history of >= 20 pack-years and if quit, quit within 15 years.
* Received referral for counseling for lung cancer screening and would qualify for LDCT.
* Health Insurance that will pay for a LDCT for lung cancer screening at either City of Hope Duarte, Newport Beach (Newport Diagnostic Imaging), or Lancaster (Renaissance Imaging/Antelope Valley Outpatient Imaging Center).
* Willingness to provide blood sample.
* English speaking.
* Consent to undergo lung cancer screening with either liquid biopsy (LB) or LDCT.

Exclusion Criteria:

* Symptoms of lung cancer.
* Chest CT scan or chest positron emission tomography (PET)/CT within 12 months.
* Any cancer diagnosis within past 5 years, excluding non-melanoma skin cancer.
* Unable to undergo LDCT at either City of Hope Duarte, Newport Beach, or Lancaster.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2029-01-28 (Estimated); Study Completion 2029-01-28 (Estimated)

PRIMARY OUTCOMES:
Screening preference | Upon completion of home liquid biopsy or LDCT, an average of 4 weeks.
  The proportion of participants who agree to undergo lung cancer screening using liquid biopsy versus LDCT, with a feasibility threshold of at least 30% preferring liquid biopsy.

SECONDARY OUTCOMES:
Participants who follow-through on screening 1 | 6 month follow-up timepoint.
  The proportion of participants who are screened with LDCT at 6 months in each screening group.
Participants who follow-through on screening 2 | 6 month follow-up timepoint.
  The proportion of participants who undergo LDCT at 6 months after receiving liquid biopsy results, stratified by test result (negative vs positive).
Participants who follow-through on screening 3 | 6 month follow-up timepoint.
  Differences in sociodemographic factors across screening preference (liquid biopsy vs. LDCT) in those who undergo screening (Exploratory).
Participants who follow-through on screening 4 | 6 month follow-up timepoint.
  Differences in sociodemographic survey scores across screening preference (liquid biopsy vs. LDCT) in those who undergo screening (Exploratory).
Participants who undergo low dose computed tomography of the chest (LDCT) after receiving liquid biopsy results | Up to 6 months
  For those who choose liquid biopsy only. Data will be summarized using counts and percentages and tested using Chi-square analysis.
Sociodemographic factors (age, sex, race/ethnicity, educational background) | At baseline visit
  Data will be summarized using means and standard deviations or counts and percentages, depending on whether the data are continuous or categorical. Univariate tests across groups will be done using t-tests (continuous) and chi-square analysis (categorical). Non-parametric tests will be used for continuous data that are non-normally distributed data (Kruskal-Wallis) and for ordinal categorical data (Jonckheere-Terpstra). Multivariable logistic regression methods will be used to determine the primary factors predicting screening preference. Data included in the model will be determined based on clinical relevance and/or significance in univariate analysis.
Survey scores across screening preference 1 | At 6 month follow up
  Survey tools will be used to understand sociodemographics, prior cancer screening, cancer worry, lung cancer risk perception, and barriers to lung cancer screening.
  Survey tools utilized:Demographics tool: including sex, race/ethnicity, education level, income.
Survey scores across screening preference 2 | At 6 month follow up
  Survey tools will be used to understand sociodemographics, prior cancer screening, cancer worry, lung cancer risk perception, and barriers to lung cancer screening.
  Survey tools utilized: Tobacco smoking history
Survey scores across screening preference 3 | At 6 month follow up
  Survey tools will be used to understand sociodemographics, prior cancer screening, cancer worry, lung cancer risk perception, and barriers to lung cancer screening.
  Survey tools utilized: Prior use of colon, breast, and lung cancer screening.
Survey scores across screening preference 4 | At 6 month follow up
  Survey tools will be used to understand sociodemographics, prior cancer screening, cancer worry, lung cancer risk perception, and barriers to lung cancer screening.
  Survey tools utilized: Lung Cancer Screening Health Beliefs Survey (lung cancer risk perception and barriers to lung cancer screening).
Survey scores across screening preference 5 | At 6 month follow up
  Survey tools will be used to understand sociodemographics, prior cancer screening, cancer worry, lung cancer risk perception, and barriers to lung cancer screening.
  Survey tools utilized: Cancer Worry Scale

CONTACTS AND LOCATIONS:
Overall Officials: Dan Raz, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States